CLINICAL TRIAL: NCT01677039
Title: An Open-label, Single-dose, Randomized, Three-way Crossover Study to Estimate the Effects of Ethanol 20% and 40% on the Bioavailability a Controlled Release Formulation of Oxycodone 20 Mg With Sequestered Naltrexone 2.4 Mg in Healthy Volunteers
Brief Title: Study to Determine the Effects of Co-Administration of Alcohol on the Absorption of Oxycodone From a Proprietary Controlled-Release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4531004
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Bioavailability; oxycodone; ethanol interaction; healthy volunteers
MeSH Terms: interventions — Water; oxycodone naltrexone combination; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator)
  Interventions: Drug: Test formulation administered with water
- Treatment B (Experimental)
  Interventions: Drug: Test formulation administered with 20% ethanol
- Treatment C (Experimental)
  Interventions: Drug: Test formulation administered with 40% ethanol

INTERVENTIONS:
Drug: Test formulation administered with water — single dose of 20 mg of test formulation with 240 mL of water
  Other Names: ALO-02 20 mg
  Arms: Treatment A
Drug: Test formulation administered with 20% ethanol — single dose of 20 mg of test formulation with 240 mL of 20% ethanol in water
  Other Names: ALO-02 20 mg
  Arms: Treatment B
Drug: Test formulation administered with 40% ethanol — single dose of 20 mg of test formulation with 240 mL of 40% ethanol
  Other Names: ALO-02 20 mg
  Arms: Treatment C

SUMMARY:
The study is designed to test whether or not the rate and extent of absorption of oxycodone from a proprietary controlled-release formulation is significantly affected by co-administration of alcohol compared with controlled conditions (when the formulation is administered with water). The primary pharmacokinetic parameters are the peak concentration of oxycodone (Cmax) and the overall exposure level of oxycodone as represented by the area under the plasma concentration-time curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* history of moderate alcohol consumption
* total body weight exceeding 64 kg

Exclusion Criteria:

* history of clinically significant disease
* history of sleep apnea
* any condition affecting drug absorption
* pregnant or nursing female subjects
* history of allergy or hypersensitivity to either oxycodone or naltrexone

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed oxycodone concentration in plasma (Cmax) | hours after dosing
Area under the oxycodone concentration versus time curve (AUC) | hours after dosing

SECONDARY OUTCOMES:
Time-to-peak concentration (Tmax) | hours after dosing
half-life of drug | hours after dosing
Vital signs and adverse events | hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Malhotra BK, Matschke K, Wang Q, Bramson C, Salageanu J. Effects of ethanol on the pharmacokinetics of extended-release oxycodone with sequestered naltrexone (ALO-02). Clin Drug Investig. 2015 Apr;35(4):267-74. doi: 10.1007/s40261-015-0278-6. PMID 25724154
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531004&StudyName=Study%20to%20Determine%20the%20Effects%20of%20Co-Administration%20of%20Alcohol%20on%20the%20Absorption%20of%20Oxycodone%20from%20a%20Proprietary%20Controlled-Release%20Formul